CLINICAL TRIAL: NCT01721876
Title: A Phase III Randomised, Double-blind, Controlled, Parallel Group Study of Intravenous Volasertib in Combination With Subcutaneous Low-dose Cytarabine vs. Placebo + Low-dose Cytarabine in Patients >=65 Years With Previously Untreated Acute Myeloid Leukaemia, Who Are Ineligible for Intensive Remission Induction Therapy
Brief Title: Volasertib in Combination With Low-dose Cytarabine in Patients Aged 65 Years and Above With Previously Untreated Acute Myeloid Leukaemia, Who Are Ineligible for Intensive Remission Induction Therapy (POLO-AML-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1230.14; 2012-002487-27 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 6727; Cytarabine

ARMS (2):
- Volasertib and Cytarabine (Experimental)
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Placebo and Cytarabine (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Cytarabine

INTERVENTIONS:
Drug: Placebo — Placebo matching Volasertib
  Arms: Placebo and Cytarabine
Drug: Volasertib — Volasertib
  Arms: Volasertib and Cytarabine
Drug: Cytarabine — Cytarabine

SUMMARY:
To investigate the efficacy, safety, and pharmacokinetics of intravenous volasertib + subcutaneous low dose cytarabine in patients >= 65 years of age with previously untreated acute myeloid leukaemia, ineligible for intensive remission induction therapy

ELIGIBILITY:
Inclusion criteria:

1. Age >= 65years.
2. Cytologically/histologically confirmed acute myeloid leukaemia (AML) according to WHO classification; (except for acute promyelocytic leukaemia (APL).
3. Previously untreated AML (except for hydroxyurea and/or corticosteroid therapy for no more than 28 days (cumulative)). Previous therapy for Myelodysplastic Syndrome (MDS) is allowed.
4. Investigator considers patient ineligible for intensive remission induction therapy based on documented medical reasons (e.g. disease characteristics like AML genetics, type of AML (de novo or secondary), and patient characteristics like performance score, concomitant diagnoses, organ dysfunctions).
5. Patient is eligible for Low-Dose Cytarabine (LDAC) treatment.
6. Eastern co-operative oncology group (ECOG) performance score <= 2 at screening.
7. Signed and dated written informed consent by start date of Screening visit in accordance with Good Clinical Practice (GCP) and local legislation.

Exclusion criteria:

1. Prior or concomitant chemotherapy for AML (with the exception of hydroxyurea and/or corticosteroid therapy for no more than 28 days (cumulative)). Please note that any prior therapy for MDS is allowed.
2. Treatment with any investigational drug within 2 weeks before first administration of present trial drug.
3. Acute promyelocytic leukaemia (French-American-British (FAB) classification subtype M3).
4. Current clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukaemic CNS involvement (no lumbar puncture required, clinical assessment per investigator´s judgement is sufficient).
5. Hypersensitivity to one of the trial drugs or the excipients.
6. Severe illness or organ dysfunction involving the heart, kidney, liver or other organ system (e.g. active infection, clinically relevant impairment of cardiac function, severe heart failure/cardiac insufficiency, unstable angina pectoris or history of recent myocardial infarction), which in the opinion of the investigator precludes treatment with LDAC.
7. Corrected QT interval according to Fridericia (QTcF) prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).The QTcF will be calculated as the mean of the 3 Electrocardiogram (ECGs) taken at screening.
8. Total bilirubin > 3 x upper limit of normal (ULN).
9. Creatinine clearance (CLcr) < 30 ml/min (estimated creatinine clearance by the Cockcroft-Gault (C-G) equation) .
10. Active hepatitis B or hepatitis C, or laboratory evidence for a chronic infection.
11. HIV infection.
12. Second malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment e.g. in prostate or breast cancer).
13. Any significant concurrent psychiatric disorder or social situation that according to the investigator´s judgement would compromise patient´s safety or compliance, interfere with consent, study participation, or interpretation of study results.
14. Known or suspected active alcohol or drug abuse.
15. Patient unable to comply with the protocol, in the opinion of the investigator.
16. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second medically acceptable method of contraception during the trial and for a minimum of 6 months after study treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 666 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (122):
- United States (4):
  - University of California, Los Angeles, California
  - St. Luke's Hospital Association of Duluth, Inc., Duluth, Minnesota
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Argentina (2):
  - Fundacion COIR, Mendoza
  - Hospital Central de Salud Zenón Santillan, San Miguel de Tucumán
- Austria (3):
  - LKH-Univ. Hospital Graz, Graz
  - LKH Leoben, Leoben
  - Hospital Hietzing, Vienna
- Belgium (8):
  - AZ Sint-Jan Brugge, Bruges
  - Brussels - UNIV Saint-Luc, Brussels
  - Haine-St-Paul - HOSP Jolimont, Haine-Saint-Paul
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Roeselare - HOSP AZ Delta, Roeselare
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Brazil (3):
  - Hospital Doutor Amaral Carvalho, Jaú
  - Hospital Mãe de Deus, Porto Alegre
  - H.C.da Fac. de Medicina de Ribeirao Preto, Ribeirão Preto
- Canada (5):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Maisonneuve-Rosemont Hospital, Montreal, Migration Data
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
- Czechia (3):
  - Hospital Hradec Kralove, Hradec Králové
  - University Hospital Plzen, Plzen-Lochotin, Plzen - Lochotin
  - Univ. Hospital Kralovske Vinohrady, Prague
- Finland (2):
  - Meilahden sairaala, Helsinki
  - TYKS, Sisätautien klinikka, Turku
- France (12):
  - HOP Amiens-Picardie Sud, Amiens
  - HOP Côte de Nacre, Caen
  - HOP Michallon, La Tronche
  - HOP André Mignot, Le Chesnay
  - HOP Dupuytren 1, Limoges
  - INS Paoli-Calmettes, Marseille
  - HOP Nantes, Hémato, Nantes, Nantes
  - HOP Saint-Antoine, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Lyon Sud, Pierre-Bénite
  - HOP Pontchaillou, Rennes
  - INS Universitaire du Cancer, Toulouse
- Germany (20):
  - Universitätsklinikum Augsburg, Augsburg
  - Med. Klinik m.S. Hämatologie und Onkologie, Berlin
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Erlangen, Erlangen
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
- Greece (5):
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Athens "Laiko", Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - University of Patras Medical School, Pátrai
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (3):
  - Semmelweis University, Budapest
  - Petz Aldar Hospital, 2nd Dept. of Internal Med., Haematology, Győr
  - Univ. of Szeged, 2nd Dept. of Internal Med., Haematology, Szeged
- India (2):
  - St. John Medical College and hospital, Bangalore
  - Tata Memorial Hospital, Mumbai
- Italy (3):
  - A.O. Spedali Civili di Brescia, Brescia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AO Città della Salute e della, Torino
- Japan (15):
  - National Hospital Organization Nagoya Medical Center, Aichi, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Akita University Hospital, Akita, Akita
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kobe University Hospital, Hyogo, Kobe
  - Tokai University Hospital, Kanagawa, Isehara
  - Yokohama City University Medical Center, Kanagawa, Yokohama
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kurashiki Central Hospital, Okayama, Kurashiki
  - Okayama University Hospital, Okayama, Okayama
  - Osaka City University Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - NTT Medical Center Tokyo, Tokyo, Sinagawa-ku
- Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Mexico
- Amsterdam UMC Locatie VUMC, Amsterdam, Netherlands
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Sykehuset Østfold Kalnes, Grålum
- Poland (2):
  - Reg. Specialist Hospital of M. Kopernik, Dept. Haematology, Lodz
  - City Hospital Torun, Department of Hematology, Torun
- Portugal (4):
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário do Porto, EPE - Hospital de Santo António, Porto
  - IPO Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar Universitário São João,EPE, Porto
- Russia (4):
  - Regional Clinical Hospital 'The Badge of Honor Order', Irkutsk
  - FSBI "N.N Blokhin Med.Res.Cent.Onc."MoH of RF, Moscow
  - Nizhniy Novgorod Reg. Clinical Hospital, Dept. Haematology, Nizhny Novgorod
  - Leningrad Reg. Clin. Hosp., Oncohematology Department No. 2, Saint Petersburg
- Netcare Pretoria East Hospital, Moreleta Park, Pretoria, South Africa
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Politècnic La Fe, Valencia
- Taiwan (3):
  - Chang-Hua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Hagege A, Ambrosetti D, Boyer J, Bozec A, Doyen J, Chamorey E, He X, Bourget I, Rousset J, Saada E, Rastoin O, Parola J, Luciano F, Cao Y, Pages G, Dufies M. The Polo-like kinase 1 inhibitor onvansertib represents a relevant treatment for head and neck squamous cell carcinoma resistant to cisplatin and radiotherapy. Theranostics. 2021 Sep 21;11(19):9571-9586. doi: 10.7150/thno.61711. eCollection 2021. PMID 34646387
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 65 years or more with previously untreated acute myeloid leukaemia, who are ineligible for intensive remission induction therapy were recruited in the phase III randomised, double-blind, placebo-controlled, parallel group study.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they (the patients) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Placebo + Low-dose Cytarabine: Patients received placebo matching to Volasertib 350 milligram (mg) intravenous infusion for 1 hour on day 1 and day 15 of each 28-day cycle, in combination with Cytarabine 20 mg subcutaneous injection given twice daily at 12 hours interval from day 1 to 10 of each 28-day cycle.
- Volasertib + Low-dose Cytarabine: Patients received Volasertib 350 mg intravenous infusion for 1 hour on day 1 and day 15 of each 28-day cycle, wherein no dose increase was allowed after a dose reduction, in combination with Cytarabine 20 mg subcutaneous injection given twice daily at 12 hours interval from day 1 to 10 of each 28-day cycle.
Period: Overall Study
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine
Started | 222 | 444
Treated | 221 | 440
Completed | 0 | 0
Not Completed | 222 | 444
Not completed — Not treated | 1 | 4
Not completed — Disease progression / relapse | 123 | 156
Not completed — Death | 6 | 13
Not completed — Adverse Event | 41 | 165
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 15 | 38
Not completed — Reason not listed | 34 | 63
Not completed — Sponsor terminated trial | 0 | 4

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all patients who had been randomised at the database snapshot.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine | Total
Number analyzed (Participants) | 222 | 444 | 666
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.5 (4.9) | 75.2 (5.4) | 75.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 203 | 290
  Male | 135 | 241 | 376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 16 | 26
  Not Hispanic or Latino | 194 | 399 | 593
  Unknown or Not Reported | 18 | 29 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 39 | 74 | 113
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 158 | 328 | 486
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 38 | 63

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: OR is the number of patients who achieved complete remission (CR) or complete remission with incomplete blood count recovery (CRi), where OR was based on the best response attained during the treatment period.
Time Frame: Response assessment was performed at the end of every 2nd cycle, (i.e. at the end of Cycle 2, 4, 6, 8, etc., and at end of treatment), i.e. up to 52 months.
Population: The randomised set (RS) included all patients who had been randomised at the database snapshot.
Measure: Number; unit: Participants
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine
Number analyzed (Participants) | 222 | 444
Participants | 38 | 123
Statistical Analysis 1: Comparison: Placebo + Low-dose Cytarabine vs Volasertib + Low-dose Cytarabine; This analysis was exploratory and descriptive; Test type: Superiority — The 2-sided test of the hypothesis was performed at a 0.05 level of significance. An odds ratio (OR) = 1 would indicate that the odds of achieving CR+CRi with Volasertib + Low-dose Cytarabine is equal to the odds of achieving CR+CRi with Placebo + Low-dose Cytarabine , whereas an OR ≠ 1 would indicate the opposite. H0, CR+CRi: OR = 1 vs. Ha, CR+CRi: OR ≠ 1; p = 0.0024, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.8751, 95% CI 2-sided [1.2432 to 2.8281] — Common odds ratio is calculated by Mantel-Haenszel estimate adjusting for the two stratification factors (baseline Eastern Cooperative Oncology Group (ECOG) and type of AML). If odds ratio is above 1 then it favours Volasertib+Low-dose Cytarabine

2. Secondary Outcome: Overall Survival (OS)
Description: OS is the key secondary endpoint and was measured from the date of randomization until death from any cause. Patients who were lost to follow-up were censored on the last date they were known to be alive.
Time Frame: From randomization until death due to any cause, up to 1557 days.
Population: RS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine
Number analyzed (Participants) | 222 | 444
Months | 6.5 [4.9 to 8.0] | 5.6 [4.5 to 6.8]
Statistical Analysis 1: Comparison: Placebo + Low-dose Cytarabine vs Volasertib + Low-dose Cytarabine; This analysis was exploratory and descriptive; Test type: Superiority — The hazard ratio (HR) between Volasertib + Low-dose Cytarabine and Placebo + Low-dose Cytarabine was tested against 1. The null hypothesis, H0,OS, was that the hazards are equal between Volasertib + Low-dose Cytarabine and Placebo + Low-dose Cytarabine, whereas the alternative hypothesis, Ha,OS, was that the hazards are not equal between the 2 treatment arms. H0, OS: HR = 1 vs. Ha, OS: HR ≠ 1; p = 0.7571, Regression, Cox — P-value is calculated from log-rank test stratified by baseline ECOG (0-1 vs. 2) and type of AML (denovo vs. secondary); Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.8 to 1.2] — Hazard ratio is calculated from Cox proportional hazard model stratified by baseline ECOG and type of AML. If hazard ratio is below 1 then it favours volasertib

3. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was measured from the date of randomisation to the date of progression or relapse, or death from any cause, whichever occurred first.
Time Frame: From randomization until disease progression or relapse or death from any cause, up to 1557 days.
Population: RS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine
Number analyzed (Participants) | 222 | 444
Months | 2.8 [2.1 to 4.9] | 3.3 [2.6 to 4.2]
Statistical Analysis 1: Comparison: Placebo + Low-dose Cytarabine vs Volasertib + Low-dose Cytarabine; This analysis was exploratory and descriptive; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6718, Regression, Cox — P-value is calculated from log-rank test stratified by baseline ECOG (0-1 vs. 2) and type of AML (denovo vs. secondary); Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.8 to 1.2] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined only for patients who achieved best overall response of CR or CRi; it was measured from the date of achievement of a remission until the date of relapse or death from any cause. Patients not known to have relapsed or died at last follow-up were censored on the date they were last examined.
Time Frame: From randomization until disease progression or relapse or death from any cause, up to 1557 days.
Population: All patients in the RS who achieved best overall response of CR or CRi.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Low-dose Cytarabine | Volasertib + Low-dose Cytarabine
Number analyzed (Participants) | 38 | 123
Months | 18.7 [11.3 to NA] — Confidence limits for the quartiles cannot be estimated due to insufficient number of participants with events. | 13.1 [6.2 to NA] — Confidence limits for the quartiles cannot be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Low-dose Cytarabine vs Volasertib + Low-dose Cytarabine; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.7 to 2.7] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after last drug administration, i.e., up to 91.4 months.
Description: The treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of Volasertib, placebo, or Low-dose Cytarabine. One patient was randomised to the Volasertib + Low-dose Cytarabine arm but only took Low-dose Cytarabine and was therefore allocated to the Placebo + Low-dose Cytarabine arm in the treated set.
Groups:
- Subjects Assigned to Placebo + Low-dose Cytarabine: Patients received placebo matching to Volasertib 350 milligram (mg) intravenous infusion for 1 hour on day 1 and day 15 of each 28-day cycle, in combination with Cytarabine 20 mg subcutaneous injection given twice daily at 12 hours interval from day 1 to 10 of each 28-day cycle.
- Subjects Assigned to Volasertib + Low-dose Cytarabine: Patients received Volasertib 350 mg intravenous infusion for 1 hour on day 1 and day 15 of each 28-day cycle, wherein no dose increase was allowed after a dose reduction, in combination with Cytarabine 20 mg subcutaneous injection given twice daily at 12 hours interval from day 1 to 10 of each 28-day cycle.
Arm/Group | Subjects Assigned to Placebo + Low-dose Cytarabine | Subjects Assigned to Volasertib + Low-dose Cytarabine
All-Cause Mortality (participants affected / at risk) | 40/222 | 138/439
Serious Adverse Events (participants affected / at risk) | 163/222 | 380/439
Other Adverse Events (participants affected / at risk) | 203/222 | 404/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Assigned to Placebo + Low-dose Cytarabine (N=222) | Subjects Assigned to Volasertib + Low-dose Cytarabine (N=439)
Anaemia (Blood and lymphatic system disorders) | 10 | 20
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 3
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 42 | 203
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 13
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 23
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 4
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 6
Atrial flutter (Cardiac disorders) | 2 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 4
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 8 | 10
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Right ventricular failure (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 8
Enteritis (Gastrointestinal disorders) | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Ileus paralytic (Gastrointestinal disorders) | 2 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Neutropenic colitis (Gastrointestinal disorders) | 0 | 5
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 6
Catheter site phlebitis (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 2
Device related thrombosis (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 2
General physical health deterioration (General disorders) | 3 | 15
Induration (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 5
Multiple organ dysfunction syndrome (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 19 | 33
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 2
Allergy to vaccine (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 3
Anal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Aspergillus infection (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 5
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 4
Bronchitis (Infections and infestations) | 1 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 3 | 12
Campylobacter sepsis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 6 | 3
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 3 | 5
Diverticulitis (Infections and infestations) | 2 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 3
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 2 | 1
Escherichia sepsis (Infections and infestations) | 0 | 4
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 3
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 1 | 2
Klebsiella infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 2
Laryngitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Lymphadenitis bacterial (Infections and infestations) | 0 | 1
Myocarditis septic (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 7
Neutropenic sepsis (Infections and infestations) | 1 | 2
Oral candidiasis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis fungal (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 44 | 113
Pneumonia fungal (Infections and infestations) | 1 | 7
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Prostatitis Escherichia coli (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 2
Pseudomonal sepsis (Infections and infestations) | 1 | 4
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 7
Respiratory tract infection fungal (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 9 | 44
Septic shock (Infections and infestations) | 10 | 28
Sinusitis (Infections and infestations) | 3 | 1
Sinusitis aspergillus (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 4
Soft tissue infection (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 3
Stenotrophomonas sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 2
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 12
Urosepsis (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 | 2
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 2
Blood pressure orthostatic decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 2
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 3
Troponin increased (Investigations) | 2 | 1
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 22
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 2 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 1 | 2
Sneddon's syndrome (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Stupor (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 4
Disorientation (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 19
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 4
Renal failure (Renal and urinary disorders) | 0 | 6
Renal impairment (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Angioplasty (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 5
Embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Large intestine infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Aortitis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Assigned to Placebo + Low-dose Cytarabine (N=222) | Subjects Assigned to Volasertib + Low-dose Cytarabine (N=439)
Anaemia (Blood and lymphatic system disorders) | 53 | 137
Febrile neutropenia (Blood and lymphatic system disorders) | 28 | 101
Leukopenia (Blood and lymphatic system disorders) | 23 | 45
Neutropenia (Blood and lymphatic system disorders) | 34 | 124
Thrombocytopenia (Blood and lymphatic system disorders) | 59 | 163
Abdominal pain (Gastrointestinal disorders) | 26 | 47
Abdominal pain upper (Gastrointestinal disorders) | 14 | 30
Constipation (Gastrointestinal disorders) | 55 | 122
Diarrhoea (Gastrointestinal disorders) | 49 | 116
Nausea (Gastrointestinal disorders) | 79 | 123
Stomatitis (Gastrointestinal disorders) | 13 | 75
Vomiting (Gastrointestinal disorders) | 27 | 71
Asthenia (General disorders) | 42 | 64
Chest pain (General disorders) | 8 | 22
Chills (General disorders) | 12 | 26
Fatigue (General disorders) | 29 | 62
Mucosal inflammation (General disorders) | 11 | 63
Oedema (General disorders) | 13 | 36
Oedema peripheral (General disorders) | 42 | 75
Pain (General disorders) | 10 | 31
Pyrexia (General disorders) | 58 | 85
Oral candidiasis (Infections and infestations) | 5 | 25
Oral herpes (Infections and infestations) | 10 | 31
Pneumonia (Infections and infestations) | 9 | 38
Urinary tract infection (Infections and infestations) | 4 | 24
Fall (Injury, poisoning and procedural complications) | 9 | 26
Alanine aminotransferase increased (Investigations) | 16 | 26
Aspartate aminotransferase increased (Investigations) | 14 | 19
Electrocardiogram QT prolonged (Investigations) | 8 | 32
Weight decreased (Investigations) | 20 | 39
Decreased appetite (Metabolism and nutrition disorders) | 43 | 82
Hyperuricaemia (Metabolism and nutrition disorders) | 13 | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 120
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 50
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 30
Dizziness (Nervous system disorders) | 18 | 43
Headache (Nervous system disorders) | 23 | 48
Insomnia (Psychiatric disorders) | 21 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 95
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 76
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 71
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 28
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 30
Petechiae (Skin and subcutaneous tissue disorders) | 24 | 73
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 27
Rash (Skin and subcutaneous tissue disorders) | 30 | 72
Haematoma (Vascular disorders) | 20 | 55
Hypertension (Vascular disorders) | 7 | 31
Hypotension (Vascular disorders) | 9 | 23
Dyspepsia (Gastrointestinal disorders) | 9 | 22
Nasopharyngitis (Infections and infestations) | 13 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 22
Confusional state (Psychiatric disorders) | 7 | 22

LIMITATIONS AND CAVEATS:
The final analysis presented in this report was conducted after 574 Overall Survival events had occurred. The final analysis was exploratory and descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.